CLINICAL TRIAL: NCT01237249
Title: A National, Open-label, Multicenter, Randomized, Comparative Phase IIb Study of Treatment for Newly Diagnosed Multiple Myeloma Patients Older Than 65 Years With Sequential Melphalan/Prednisone/Velcade (MPV) Followed by Revlimid/Low Dose Dexamethasone (Rd) Versus Alternating Velcade/Melphalan/Prednisone (MPV) With Revlimid/Low Dose Dexamethasone (Rd).
Brief Title: Study of Treatment for Newly Diagnosed Multiple Myeloma Patients Older Than 65 Years With Sequential Melphalan/Prednisone/Velcade (MPV) Followed by Revlimid/Low Dose Dexamethasone (Rd) Versus Alternating Velcade/Melphalan/Prednisone (MPV) With Revlimid/Low Dose Dexamethasone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Janssen-Cilag Ltd. (Industry); Celgene (Industry); TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM2010MAS65
Record Dates: First submitted 2010-11-04; First posted 2010-11-09 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Velcade; Revlimid
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Prednisone; Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPV followed by Revlimid/Low Dose Dexamethasone (Rd) (Active Comparator): Melphalan/Prednisone/Velcade (MPV) followed by Revlimid/Low Dose Dexamethasone (Rd)
  Interventions: Drug: Melphalan; Drug: Prednisone; Drug: Velcade
- Alternating MPV with Revlimid/Low Dose Dexamethasone (Experimental): Alternating Velcade/Melphalan/Prednisone (MPV) with Revlimid/Low Dose Dexamethasone (Rd)
  Interventions: Drug: Revlimid; Drug: Dexamethasone

INTERVENTIONS:
Drug: Melphalan
  Arms: MPV followed by Revlimid/Low Dose Dexamethasone (Rd)
Drug: Prednisone
  Arms: MPV followed by Revlimid/Low Dose Dexamethasone (Rd)
Drug: Velcade
  Arms: MPV followed by Revlimid/Low Dose Dexamethasone (Rd)
Drug: Revlimid
  Arms: Alternating MPV with Revlimid/Low Dose Dexamethasone
Drug: Dexamethasone
  Arms: Alternating MPV with Revlimid/Low Dose Dexamethasone

SUMMARY:
This is a national, multicenter, open-label, randomized, comparative study designed to compare, first, the TTP of the two treatment schemes proposed (MPV followed by Rd or MPV alternating with Rd) in newly diagnosed MM patients older than 65 years. This comparison will be performing in terms of both efficacy and safety. Up to 120 patients will be included in each treatment arm and evaluated at scheduled visits in up to 3 study periods: Pre-treatment, Treatment and Follow-up.

Primary outcome measure:

* To evaluate the efficacy in terms of time to progression (TTP) at 18 months of MPV and Rd used as either in a sequential or alternating approach in newly diagnosed MM patients older than 65 years.
* To evaluate the toxicity (safety and tolerability) of the sequential versus the alternating use of MPV and Rd.

Secondary outcome measure:

* To evaluate the response, duration of response, progression free survival (PFS), time to next therapy (TNT) and overall survival (OS) in the two different groups of patients.
* To identify, within the group of patients treated with the alternating scheme, the biological characteristics (including a comprehensive genomic analysis) of those patients resistant to one or the other, and patients refractory to both treatments

DETAILED DESCRIPTION:
The Pre-treatment period includes Screening visit. After providing written informed consent form to participate in the study, patients will be evaluated for eligibility during a screening period of 14 days (Days -14 to -1). If patients meet all inclusion and exclusion criteria will be randomized at the moment of entry in the trial in a 1:1 allocation to receive either MPV followed by Rd (Treatment Group A) or MPV alternating with Rd (Treatment Group B).

Patients in the Treatment Group A will receive nine cycles of MPV consisting on one 6-weeks cycle of Velcade (Bortezomib) as an intravenous bolus twice weekly (days 1, 4, 8, 11, 22, 25, 29 and 32) followed by a 10 day rest period (day 33 to 42), in combination with oral Melphalan, once daily on days 1 to 4 and oral Prednisone, once daily on days 1 to 4, followed by eight 4-weeks cycles of Velcade (Bortezomib) as an intravenous bolus on days 1, 8, 15 and 22 followed by a 6 day rest period (days 23 to 28), in combination with Melphalan and Prednisone per os once daily on days 1 to 4, followed by a 24-day rest period (days 5 to 28). After the nine MPV cycles, patients will receive nine cycles of Rd consisting on 4-weeks cycles, including Revlimid (lenalidomide), once daily on days 1-21 followed by a 7 day rest period (days 22 to 28) plus oral dexamethasone, once weekly on days 1,8,15 and 22, followed by a 6 day rest period (days 23 to 28).

Patients in the Treatment Group B will receive the same schedule of therapy, but the MPV cycles will be alternated with Rd cycles. In this treatment Group B, patients will be again randomized to start receiving either MPV or Rd as first cycle of therapy. Overall, patients will receive an identical number of cycles, nine cycles of MPV and nine of Rd. Patients randomized to Treatment Group A relapsing/progressing or with major toxicities under treatment with MPV will be crossover to receive Rd, but only after study coordinator approval.

During the Treatment Period, patients will be evaluated at day 1 of each cycle. After completion of the Treatment Period, all patients will be evaluated every 2 months thereafter.

Safety will be assessed by the monitoring of adverse events, physical examinations, vital signs measurements, and haematology and clinical chemistry test. Response to treatment will be based on EBMT an IMWG criteria. Response to treatment will be evaluated at day 1 of each induction cycle, and every 2 months during thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before starting any study-specific procedure.
2. Symptomatic elderly MM newly diagnosed by EBMT criteria older than 65 years.
3. Performance status (ECOG) ≤ 2.
4. Have pre-treatment clinical laboratory values meeting the following criteria within 14 days of randomization:

   * platelet count ≥ 75x109/L
   * haemoglobin ≥ 8g/dL
   * absolute neutrophil count (ANC) ≥ 1.0x109/L
   * Serum bilirubin ≤ 1.5 mg/dL and alkaline phosphatise ≤ 2.5 x ULN AST, ALT ≤ 2.5 x ULN
   * Serum creatinine ≤2,5 mg/dl

Exclusion Criteria:

1. Patient previously received treatment with Velcade or Revlimid.
2. Patient previously received treatment for Multiple Myeloma.
3. Patient has ≥ Grade 2 peripheral neuropathy within 14 days before enrolment.
4. Patient has hypersensitivity to bortezomib, boron, mannitol or lenalidomide.
5. Patient has received other investigational drugs with 28 days before enrolment.
6. Patient had a myocardial infarction within 6 months of enrolment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
7. Patient currently is enrolled in another clinical research study and/or is receiving an investigational agent for any reason.
8. Radiation therapy within 30 days before randomization, at least patient has had antialgic radiation. Radiation therapy will be afterwards permitted during the treatment period if it is indicated due to the presence of plasmacytomas

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-02; Primary Completion 2014-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy in terms of time to progression (TTP) at 18 months of MPV and Rd used as either in a sequential or alternating approach in newly diagnosed MM patients older than 65 years. | 18 months
To evaluate the toxicity (safety and tolerability) of the sequential versus the alternating use of MPV and Rd,in terms of adverse events presented in both groups of patients | 6 months

SECONDARY OUTCOMES:
To evaluate the response in both groups of patients | 1 year
To identify, within the group of patients treated with the alternating scheme, the biological characteristics (including a comprehensive genomic analysis) of those patients resistant to one or the other, and patients refractory to both treatments | 2 years
Duration of response in two groups of patients | 2 years
Progression free survival (PFS) in two different groups of patients | 18 months
Time to next therapy (TNT) | 2 years
Overall survival (OS) in the two different groups of patients | 5 years

CONTACTS AND LOCATIONS:
Locations (63):
- Spain (63):
  - H. Son Llatzer, Palma de Mallorca, Balearic Islands
  - H. Vall d'Hebron, Barcelona, Barcelona, Barcelona
  - ICO - Duran i Reynals, Hospitalet de Llobregat, Barcelona, Barcelona
  - Hospital General de Castellón, Castellon, Castellón
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Joan XXIII, Tarragona, Tarragona
  - Hospital Universitario Dr. Peset, Valencia, Valencia
  - Miguel Servet, Zaragoza, Zaragoza
  - Fundación Hospital Alcorcón, Alcorcón
  - Hospital de Badalona Germans Trias i Pujol, Badalona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital Puerta del Mar, Cadiz
  - Complejo Hospitalario de Cáceres, Cáceres
  - Hospital General, Ciudad Real
  - Hospital Virgen de la Luz, Cuenca
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Francesc Borja, Gandia
  - ICO - Josep Trueta, Girona
  - Hospital General de Guadalajara, Guadalajara
  - H. de Jerez, Jerez de la Frontera
  - Complejo Hospitalario León, León
  - Clínica Puerta de Hierro, Madrid
  - Hospital 12 de Octubre. Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital de Fuenlabrada, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital de Madrid, S.A.- Norte Hospital General, Madrid
  - Hospital del Tajo, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Infanta Sofia, Madrid
  - Hospital la Paz, Madrid
  - Hospital Severo Ochoa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - MD Anderson, Madrid
  - Althaia, Manresa
  - Complejo Hospital Costa del Sol, Málaga
  - Hospital Nuestra Señora de Valme, Málaga
  - Hospital General Univeristario Morales Messeguer, Murcia
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital de la Diputación de Navarra, Navarra
  - Hospital de Gran Canaria Doctor Negrín, Palma de Gran Canaria
  - Complejo Asistencial Son Dureta, Palma de Mallorca
  - Hospital Virgen del Camino, Pamplona
  - Corporació Sanitaria Parc Taulí, Sabadell
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hoaspital Marqués de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Complejo Hospitalario Regional Virgen del Rocío, Seville
  - Hospital Nuestra Señora del Prado, Toledo
  - Hospital Virgen de la Salud, Toledo
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clínico de Valencia., Valencia
  - Hospital La Fe, Valencia
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital Virgen de la Concha, Zamora
  - Hospital Clinico Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Quwaider D, Corchete LA, Misiewicz-Krzeminska I, Sarasquete ME, Perez JJ, Krzeminski P, Puig N, Mateos MV, Garcia-Sanz R, Herrero AB, Gutierrez NC. DEPTOR maintains plasma cell differentiation and favorably affects prognosis in multiple myeloma. J Hematol Oncol. 2017 Apr 18;10(1):92. doi: 10.1186/s13045-017-0461-8. PMID 28420429
- [Derived] Paiva B, Cedena MT, Puig N, Arana P, Vidriales MB, Cordon L, Flores-Montero J, Gutierrez NC, Martin-Ramos ML, Martinez-Lopez J, Ocio EM, Hernandez MT, Teruel AI, Rosinol L, Echeveste MA, Martinez R, Gironella M, Oriol A, Cabrera C, Martin J, Bargay J, Encinas C, Gonzalez Y, Van Dongen JJ, Orfao A, Blade J, Mateos MV, Lahuerta JJ, San Miguel JF; Grupo Espanol de Mieloma/Programa para el Estudio de la Terapeutica en Hemopatias Malignas (GEM/PETHEMA) Cooperative Study Groups. Minimal residual disease monitoring and immune profiling in multiple myeloma in elderly patients. Blood. 2016 Jun 23;127(25):3165-74. doi: 10.1182/blood-2016-03-705319. Epub 2016 Apr 26. PMID 27118453
- [Derived] Paiva B, Corchete LA, Vidriales MB, Puig N, Maiso P, Rodriguez I, Alignani D, Burgos L, Sanchez ML, Barcena P, Echeveste MA, Hernandez MT, Garcia-Sanz R, Ocio EM, Oriol A, Gironella M, Palomera L, De Arriba F, Gonzalez Y, Johnson SK, Epstein J, Barlogie B, Lahuerta JJ, Blade J, Orfao A, Mateos MV, San Miguel JF; Spanish Myeloma Group / Program for the Study of Malignant Blood Diseases Therapeutics (GEM / PETHEMA) Cooperative Study Groups. Phenotypic and genomic analysis of multiple myeloma minimal residual disease tumor cells: a new model to understand chemoresistance. Blood. 2016 Apr 14;127(15):1896-906. doi: 10.1182/blood-2015-08-665679. Epub 2016 Jan 11. PMID 26755711
- See also: Spanish Association of Hematology — http://aehh.org